CLINICAL TRIAL: NCT00447122
Title: BrUOG-PA-209: Lapatinib and Gemcitabine for Metastatic Pancreaticobiliary Cancer: A Phase I Study #108181
Brief Title: BrUOG-PA-209: Lapatinib and Gemcitabine for Metastatic Pancreaticobiliary Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow enrollment and lack of funding
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Memorial Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-PA-209
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Lapatinib; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- treatment 1 (Experimental): Gemcitabine 1000mg/m2 with lapatinib 1000mg/d weekly x 3 weeks
  Interventions: Drug: Gemcitabine 1000mg/m2 30 minutes; Drug: Lapatinib 1000mg/d
- treatment 2 (Experimental): Gemcitabine 1000mg/m2 with lapatinib 1500mg/d weekly X 3 weeks
  Interventions: Drug: Gemcitabine 1000mg/m2 30 minutes; Drug: Lapatinib 1500mg/d
- treatment 3 (Experimental): gemcitabine 1000 mg/m2 and oxaliplatin 100 mg/m2 on days 1 and 14 of a 28-day cycle with lapatinib 1000 mg/d
  Interventions: Drug: Lapatinib 1000mg/d; Drug: Gemcitabine 1000mg/m2 100minutes; Drug: Oxaliplatin 100mg/m2
- treatment 4 (Experimental): gemcitabine 1000 mg/m2 and oxaliplatin 100 mg/m2 on days 1 and 14 of a 28-day cycle with lapatinib 1500 mg/d
  Interventions: Drug: Lapatinib 1500mg/d; Drug: Gemcitabine 1000mg/m2 100minutes; Drug: Oxaliplatin 100mg/m2

INTERVENTIONS:
Drug: Gemcitabine 1000mg/m2 30 minutes — 1000mg/m2 30 minutes
  Other Names: Gemzar
  Arms: treatment 1; treatment 2
Drug: Lapatinib 1000mg/d — 1000mg/d
  Other Names: Tykerb; Tyverb
  Arms: treatment 1; treatment 3
Drug: Lapatinib 1500mg/d — 1500mg/d
  Other Names: Tykerb; Tyverb
  Arms: treatment 2; treatment 4
Drug: Gemcitabine 1000mg/m2 100minutes — 1000mg/m2 100minutes
  Other Names: Gemzar
  Arms: treatment 3; treatment 4
Drug: Oxaliplatin 100mg/m2 — 100mg/m2
  Other Names: Eloxatin
  Arms: treatment 3; treatment 4

SUMMARY:
Phase I study of lapatinib and gemcitabine for patients with metastatic pancreaticobiliary cancer.

DETAILED DESCRIPTION:
To evaluate the safety/tolerability and potential antitumor activity of lapatinib, at dose ranges of 1000 to 1500 mg/d, in combination with gemcitabine and gemcitabine/oxaliplatin (GEMOX) in patients with advanced pancreaticobiliary cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to have histologically or pathologically confirmed, metastatic adenocarcinoma of the pancreas
* No prior chemotherapy for pancreatic cancer.
* ECOG performance status 0-1
* Must retain ability to swallow oral medications
* Age > 18. Because no dosing or adverse event data are currently available on the use of lapatinib in patients < 18 years of age, children are excluded from this study.
* Women of child bearing potential must be non pregnant and non lactating.The effects of lapatinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female is eligible to enter and participate in the study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:

    * Has had a hysterectomy,
    * Has had a bilateral oophorectomy (ovariectomy),
    * Has had a bilateral tubal ligation, or
    * Is post-menopausal(demonstration of total cessation of menses for ³1 year).
  * Childbearing potential, has a negative serum pregnancy test within 2 weeks prior to treatment to rule out pregnancy.
  * Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment.

    * Intrauterine Device (IUD),
    * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
    * Complete abstinence from sexual intercourse for two weeks before exposure to investigational products, throughout the clinical trial, and for at least one week after the last dose of investigational product.
    * Double barrier contraception (condom with spermicidal jelly, foam, suppository, or film; diaphragm with spermicide; or male condom and diaphragm).
    * Vasectomy
* Adequate hematologic function: ANC ≥ 1500/ul, platelets ≥ 100,000/ul. Adequate hepatic function with total bilirubin ≤ 2.0 mg/dL and ALT or AST ≤ 2x ULN. (Patients with liver metastases may have AST/ALT less than or equal to 5x upper limit of normal).
* Adequate renal function: creatinine ≤ 2.0 mg/dL
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan. Note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution.
* Life expectancy of at least 12 weeks
* Signed informed consent

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Prior treatment with lapatinib or any EGFR targeting therapies.
* Prior treatment with systemic chemotherapy for pancreatic cancer.
* Clinical evidence of brain metastases or leptomeningeal disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active cardiac disease, defined as:

  * History of uncontrolled angina
  * Myocardial infarction < 6 months from study entry
  * Uncontrolled or symptomatic congestive heart failure
  * Ejection fraction below the institutional normal limit
  * Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* The subject has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib
* Participation in any investigational study within 28 days prior to study enrolment
* Any major surgery (insertion of a vascular access device or laparoscopy is not considered a major surgery), within the last 4 weeks.
* Pregnant or lactating females are excluded from this study because lapatinib is member of the 4-anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lapatinib, breastfeeding should be discontinued if the mother is treated with lapatinib.
* Uncontrolled malabsorption syndrome significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption of lapatinib.
* Any unresolved bowel obstruction.
* The patient has inadequate venous access in the clinical judgment of the investigator or designated clinical staff.
* Patient is taking any medication on the prohibited medications list in
* Patients requiring oral anticoagulants (coumadin, warfarin) are eligible provided there is increased vigilance with respect to monitoring INR. If medically appropriate and treatment available, the investigator may also consider switching these patients to LMW heparin, where an interaction with lapatinib is not expected.
* Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (1):
- Lifespan Hospitals, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 patients were enrolled
Groups:
- Arm 1: lapatinib, 1,000 mg/day, and Gemcitabine, 1000mg/m2
- Arm 2: Gem 1000mg/m2, lapatinib 1500mg/d
- Arm 3: Gem 1000mg/m2 100 minutes oxaliplatin 100mg/m2 lapatinib 1000mg/d
- Arm 4: Gem 1000mg/m2 100 minutes oxaliplatin 100mg/m2 lapatinib 1500mg/d
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 3 | 11 | 6 | 5
Completed | 3 | 10 | 6 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — worsening medical condition -came off | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Gemcitabine, 1000mg/m2 and lapatinib 1000mg/d
- Arm 2: Gemcitabine, 1000mg/m2 and lapatinib 1500mg/d
- Arm 3: Gemcitabine, 1000mg/m2 over 100minutes lapatinib 1000mg/d oxaliplatin 100mg/m2
- Arm 4: Gemcitabine, 1000mg/m2 over 100minutes lapatinib 1500mg/d oxaliplatin 100mg/m2
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 3 | 11 | 6 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 6 | 5 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 4 | 4 | 18
  Male | 1 | 3 | 2 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 11 | 6 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival for Patients With Metastatic Pancreatic Cancer.
Time Frame: Date of study entry until the date of death, up to 12 months.
Measure: Number; unit: participants
Groups:
- Arm 1: Gem 1000mg/m2 lapatinib 1000mg/d
- Arm 2: Gem 1000mg/m2 lapatinib 1500mg/d
- Arm 3: Gem 1000mg/m2 lapatinib 1000mg/d oxaliplatin 100mg/m2
- Arm 4: Gem 1000mg/m2 lapatinib 1500mg/d oxaliplatin 100mg/m2
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 3 | 11 | 6 | 5
participants | 3 | 10 | 6 | 5

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/11 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/11 | 1/6 | 2/5
Other Adverse Events (participants affected / at risk) | 0/3 | 1/11 | 1/6 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=3) | Arm 2 (N=11) | Arm 3 (N=6) | Arm 4 (N=5)
pneumocystis sepsis and ARDS (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=3) | Arm 2 (N=11) | Arm 3 (N=6) | Arm 4 (N=5)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (11) | 0 (0) | 0 (0)
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)

LIMITATIONS AND CAVEATS:
Early termination due to slow enrollment and lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No